CLINICAL TRIAL: NCT01586754
Title: Subclinical Organ Damage in Overweight and Obese Patients: Does Presence of Metabolic Syndrome Matter?
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Goztepe Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Esra Ekiz, Medical Doctor/Resident, Goztepe Training and Research Hospital
Other Study IDs: 34
Record Dates: First submitted 2012-04-25; First posted 2012-04-27 (Estimated); Last update posted 2012-04-27 (Estimated); Status verified 2012-04

CONDITIONS: Metabolic Syndrome; Subclinical Organ Damage; Overweight; Obese
Keywords: metabolic syndrome; obesity; endothelial damage; homocysteine; microalbumin; carotis intima-media thickness
MeSH Terms: conditions — Metabolic Syndrome; Overweight; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood will be drawn from patients for routine biochemical analyses for glucose, urea, creatinine, liver function tests, thyroid function tests, electrolytes and homocysteine and also glucose tolerance test. Spot urine samples will be drawn for assessment of microalbuminuria.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- With Metabolic Syndrome
- Without Metabolic Syndrome

SUMMARY:
Microalbuminuria and homocysteine levels are shown to be markers for endothelial dysfunction and subclinical organ damage and predictors of cardiovascular risk in several epidemiologic and randomized clinical trials. Carotis intima-media thickness is also found to be elevated in early stages of atherosclerosis. Recent studies have shown correlations between homocysteine, microalbumin levels and carotis intima-media thickness in type 2 diabetics but no data exists for obese or overweight patients who also have metabolic syndrome, in terms of markers of subclinical organ damage. Since obesity is a risk factor for cardiovascular disease and since it is known that patients with metabolic syndrome are at higher risk of cardiovascular events, the investigators wanted to examine whether there is an association between homocysteine, microalbumin levels and carotid intima-media thickness in patients with or without metabolic syndrome, who are either overweight or obese.

ELIGIBILITY:
Inclusion Criteria:

1. 18-80 years
2. BMI >= 25
3. Ex or non-smokers (must have quit smoking at least 5 years ago)

Exclusion Criteria:

1. NIDDM or IDDDM
2. Nephropathy (GFR < 60 ml/min), previous history of coronary artery disease or peripheral arterial disease
3. Current smokers
4. Active infection or other acute illness

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Obese or overweight patients, aged between 18-80 who are non-smokers, with a GFR > 60 ml/min and without any history of diabetes (insulin dependent or non-insulin dependent), coronary artery disease or peripheral arterial disease, attending to hyperlipidemia and obesity outpatient clinic.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2011-10; Primary Completion 2012-04 (Estimated); Study Completion 2012-05 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: ESRA EKIZ, MD, Principal Investigator — Istanbul Medeniyet University Goztepe Training and Research Hospital
Locations (1):
- Istanbul Medeniyet University Goztepe Training and Research Hospital, Istanbul, Turkey (Türkiye)